CLINICAL TRIAL: NCT03257605
Title: Implementation of a Pharmacist-Led Pharmacogenomics Service for the Program of All-inclusive Care for the Elderly (PHARM-GENOME-PACE)
Brief Title: A Pharmacist Implemented Pharmacogenomics Service in the Program of All-inclusive Care for the Elderly
Acronym: PACE
Status: Completed | Type: Observational
Sponsor: Tabula Rasa HealthCare (Industry)
Collaborators: Coriell Life Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHARM-GENOME-PACE 1173
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pharmacogenomics; Medication Therapy Management
Keywords: Pharmacogenomics; Medication Therapy Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Participants enrolled in PACE who underwent pharmacogenomics testing as part of their medical care and also consented to the use of their de-identified data for research purposes.

SUMMARY:
The aim of this study is to evaluate and describe the feasibility of implementing a pharmacist-led pharmacogenomics service for the Program of All-inclusive Care for the Elderly (PACE), a community-based practice setting.

DETAILED DESCRIPTION:
To determine if a pharmacogenomics (PGx) service can become a component of everyday practice, feasibility assessments are needed. While some researchers have begun to assess the feasibility of implementing PGx into pharmacy practice in community-based practice settings, none that we are aware have assessed such feasibility for the Program of All-inclusive Care for the Elderly (PACE). The primary objective of this feasibility study is to evaluate the processes that were involved in implementing a pharmacist-led PGx service for PACE and to describe process-related challenges and solutions associated with implementation. Secondary objectives include: describe pharmacists' roles in the implementation process; report aggregate PGx test results, including genetic variants and drug-gene interactions; and describe pharmacists' recommendations to personalize drug regimens for PACE participants and prescribers' acceptance of these recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Participant enrolled in PACE contractually receiving pharmacy services from Tabula Rasa Healthcare (CareKinesis Pharmacy) during the project time period (May 2014 through June 2016); and
* PACE prescriber ordered a pharmacogenomics test for the participant as part of clinical care; and,
* PACE participant consented to a pharmacogenomics test; and,
* CareKinesis pharmacist provided a consultation directly to PACE prescriber based on the participant's pharmacogenomics test results.

Exclusion Criteria:

* Participant dis-enrolled from PACE prior to receiving pharmacogenomics test results and/or prior to CareKinesis pharmacist providing consultative services; or,
* Participant did not complete the pharmacogenomics test.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the United States, PACE is a medical home model for participants >=55 years of age who are certified by their state as needing nursing-facility level of care but can reside safely in the community through PACE, as an alternative to institutionalization. Participants enrolled in PACE who underwent pharmacogenomics testing as part of their medical care and also consented to the use of their de-identified data for research purposes were eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Implementation Primary | 24 months
  Qualitative description of process-related challenges and successes as assessed by observation

SECONDARY OUTCOMES:
Implementation Secondary | 24 months
  Qualitative description of pharmacists' roles as assessed by observation
Pharmacogenomic Testing | 24 months
  Quantitative description of pharmacogenomic testing results as assessed by analysis of genotype and phenotype
Pharmacist Recommendations | 24 months
  Qualitative and quantitative descriptions of pharmacists' pharmacogenomic-based recommendations to prescribers as assessed by evaluation of consultations
Prescriber Acceptances | 24 months
  Qualitative and quantitative descriptions of prescribers' acceptances of pharmacists' recommendations as assessed by responses and post-consultation drug profile reviews

CONTACTS AND LOCATIONS:
Overall Officials: Kevin T Bain, PharmD, MPH, Principal Investigator — Tabula Rasa HealthCare

IPD SHARING:
Plan to Share IPD: No
Information about participants' drugs will not be shared with either the laboratory company or laboratory interpretive company. There will be no disclosure of participant information and no details of participant identity will be part of any presentation or publication of the research. Participant confidentiality will be held in strict trust by the project investigators. This confidentiality extends to any participation-related information as well as biological samples and PGx test results. The project data or other information generated will be held in strict confidence. No information concerning the project or the data will be released to any unauthorized third party without prior written consent.

REFERENCES:
- [Background] Evans WE, McLeod HL. Pharmacogenomics--drug disposition, drug targets, and side effects. N Engl J Med. 2003 Feb 6;348(6):538-49. doi: 10.1056/NEJMra020526. No abstract available. PMID 12571262
- [Background] Hocum BT, White JR Jr, Heck JW, Thirumaran RK, Moyer N, Newman R, Ashcraft K. Cytochrome P-450 gene and drug interaction analysis in patients referred for pharmacogenetic testing. Am J Health Syst Pharm. 2016 Jan 15;73(2):61-7. doi: 10.2146/ajhp150273. PMID 26721535
- [Background] Evans WE, Johnson JA. Pharmacogenomics: the inherited basis for interindividual differences in drug response. Annu Rev Genomics Hum Genet. 2001;2:9-39. doi: 10.1146/annurev.genom.2.1.9. PMID 11701642
- [Background] Tannenbaum C, Sheehan NL. Understanding and preventing drug-drug and drug-gene interactions. Expert Rev Clin Pharmacol. 2014 Jul;7(4):533-44. doi: 10.1586/17512433.2014.910111. Epub 2014 Apr 19. PMID 24745854
- [Background] Ferreri SP, Greco AJ, Michaels NM, O'Connor SK, Chater RW, Viera AJ, Faruki H, McLeod HL, Roederer MW. Implementation of a pharmacogenomics service in a community pharmacy. J Am Pharm Assoc (2003). 2014 Mar-Apr;54(2):172-80. doi: 10.1331/JAPhA.2014.13033. PMID 24632932
- [Background] Haga SB, LaPointe NM, Cho A, Reed SD, Mills R, Moaddeb J, Ginsburg GS. Pilot study of pharmacist-assisted delivery of pharmacogenetic testing in a primary care setting. Pharmacogenomics. 2014 Sep;15(13):1677-86. doi: 10.2217/pgs.14.109. PMID 25410893
- [Background] Haga SB, Allen LaPointe NM, Moaddeb J, Mills R, Patel M, Kraus WE. Pilot study: incorporation of pharmacogenetic testing in medication therapy management services. Pharmacogenomics. 2014 Nov;15(14):1729-1737. doi: 10.2217/pgs.14.118. PMID 25493566
- [Background] Moaddeb J, Mills R, Haga SB. Community pharmacists' experience with pharmacogenetic testing. J Am Pharm Assoc (2003). 2015 Nov-Dec;55(6):587-594. doi: 10.1331/JAPhA.2015.15017. PMID 26409205
- [Background] Welch BM, Kawamoto K. Clinical decision support for genetically guided personalized medicine: a systematic review. J Am Med Inform Assoc. 2013 Mar-Apr;20(2):388-400. doi: 10.1136/amiajnl-2012-000892. Epub 2012 Aug 25. PMID 22922173
- [Derived] Bain KT, Knowlton CH, Matos A. Cost avoidance related to a pharmacist-led pharmacogenomics service for the Program of All-inclusive Care for the Elderly. Pharmacogenomics. 2020 Jul;21(10):651-661. doi: 10.2217/pgs-2019-0197. Epub 2020 Jun 9. PMID 32515286
- [Derived] Bain KT, Matos A, Knowlton CH, McGain D. Genetic variants and interactions from a pharmacist-led pharmacogenomics service for PACE. Pharmacogenomics. 2019 Jul;20(10):709-718. doi: 10.2217/pgs-2019-0047. Epub 2019 Aug 1. PMID 31368837